CLINICAL TRIAL: NCT06338189
Title: The 5Ad Diet for Functional Bowel Disorders: A Randomised Controlled Trial Against the Low FODMAP Diet
Brief Title: The 5Ad Diet for Functional Bowel Disorders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Suffolk (Other)
Responsible Party: Principal Investigator, Camilla Bunn, Principal Investigator, University of Suffolk
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: USuffolk
Record Dates: First submitted 2024-03-15; First posted 2024-03-29 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Functional Bowel Disorder; Irritable Bowel Syndrome; Food Intolerance; Food Intolerance Syndromes
Keywords: The 5Ad Diet; The Low FODMAP Diet; Irritable Bowel Syndrome; Functional Constipation; Functional Diarrhoea; Functional Bloating
MeSH Terms: conditions — Irritable Bowel Syndrome; Food Intolerance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The 5Ad Diet (Active Comparator): Participants are required to follow the 5Ad diet for 7 days, followed by a washout phase for 7 days, before crossing over to the active phase of the low FODMAP diet for 7 days.
  Interventions: Other: The 5Ad Diet; Other: The Low FODMAP Diet
- The Low FODMAP Diet (Active Comparator): Participants are required to follow the active phase of the low FODMAP diet for 7 days, followed by a washout phase for 7 days, before crossing over to the 5Ad diet for 7 days.
  Interventions: Other: The 5Ad Diet; Other: The Low FODMAP Diet

INTERVENTIONS:
Other: The 5Ad Diet — Participants are to follow the 5Ad diet.
Other: The Low FODMAP Diet — Participants are to follow the active phase of the Low FODMAP diet.

SUMMARY:
The goal of this randomised controlled trial (RCT) is to compare the efficacy of the newly developed 5Ad diet against the widely researched low fermentable oligo-, di-, monosaccharide and polyols (FODMAP) diet in reducing gastrointestinal symptoms associated with functional bowel disorders/food intolerances.

The primary aims of this RCT are to determine:

* Whether the 5Ad diet is at least as effective as the low FODMAP diet in reducing gastrointestinal symptoms associated with FBDs/food intolerances.
* Whether either the 5Ad diet or the low FODMAP diet are effective in reducing mental and physical fatigue.

To achieve the above aims, an RCT will be conducted with the 5Ad diet in one arm vs the active phase of the low FODMAP diet in the other arm, in a cross-over design with a 7 days washout phase in between. Both dietary protocols will be followed by each participant for 7 days.

Researchers will compare the results from the 2 dietary protocols in order to ascertain the superiority of one over the other in regards to 6 gastrointestinal symptoms (abdominal pain, bloating, flatulence, bowel urgency, straining and incomplete defecation), stool form and frequency of defecation.

DETAILED DESCRIPTION:
Functional Bowel Disorders (FBDs) are characterised by chronic gastrointestinal symptoms including abdominal pain, constipation, bloating, diarrhoea, alternating abdominal symptoms, and irregular frequency of bowel movements among others in the absence of any intestinal abnormality. The prevalence of FBDs ranges from 15 - 20% worldwide, with remarkable economic burden on health systems and significant impact on the quality of life of sufferers. It is estimated that between 60% - 89% of individuals that suffer from FBDs find that foods exacerbate their symptoms. Therefore, dietary therapies are frequently implemented to assist with symptom relief in these individuals.

Although the low FODMAP diet is the most commonly followed diet for the treatment of FBDs, there are concerns regarding it's complexity, restrictiveness, nutritional adequacy, and effectiveness. Therefore, the 5Ad diet was designed to fill a gap in the existing research and to overcome the limitations associated with existing dietary approaches.

Preliminary findings from the first study in 2019 suggested that the 5Ad diet might be a promising universal approach for varying forms and severities of FBDs. Therefore, an RCT is needed to substantiate these previous results. Thus, this RCT aims to determine whether the 5Ad diet is at least as effective as the low FODMAP diet in reducing gastrointestinal symptoms associated with FBDs/food intolerances.

ELIGIBILITY:
Inclusion Criteria:

Individuals are eligible for the study if all of the following criteria are met:

* Suffers chronically from either constipation, diarrhoea, or an alternation of both, bloating, flatulence or abdominal pain, incomplete defecation, straining and bowel urgency.
* Symptoms must be present for ≥ 2 times per week, with symptom onset occurring at least 3 months prior to participation.
* Participants taking prescribed medications which may affect bowel function are included only if the intake is maintained throughout the entire intervention period.

Exclusion Criteria:

Individuals are excluded from the study if any of the following criteria are met:

* Pregnant.
* Known underlying pathology (e.g., Crohn's disease, ulcerative colitis, celiac disease).
* History of abdominal/gastrointestinal surgery within 1 year prior to participation.
* History of antibiotic use in the last 6 weeks prior to participation.
* Allergic to the foods specified in both the 5Ad diet and the low FODMAP diet.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2022-05-08 (Actual); Primary Completion 2025-04-01 (Actual); Study Completion 2025-04-01 (Actual)

PRIMARY OUTCOMES:
Abdominal Pain | Assessed daily throughout both dietary protocols (7 days for each dietary protocol)
  Abdominal pain will be recorded daily in a symptom diary and measured using a 4 point Likert-type scale, coded from 0 - 10 for conversion into continuous variables (None = 0; Mild = 1 - 3; Moderate = 4 - 6 ; Severe = 7 - 10).
Abdominal Bloating | Assessed daily throughout both dietary protocols (7 days for each dietary protocol)
  Abdominal bloating will be recorded daily in a symptom diary and measured using a 4 point Likert-type scale, coded from 0 - 10 for conversion into continuous variables (None = 0; Mild = 1 - 3; Moderate = 4 - 6 ; Severe = 7 - 10).
Flatulence | Assessed daily throughout both dietary protocols (7 days for each dietary protocol)
  Flatulence will be recorded daily in a symptom diary and measured using a 4 point Likert-type scale, coded from 0 - 10 for conversion into continuous variables (None = 0; Mild = 1 - 3; Moderate = 4 - 6 ; Severe = 7 - 10).
Bowel Urgency | Assessed daily throughout both dietary protocols (7 days for each dietary protocol)
  Bowel urgency will be recorded daily in a symptom diary and measured using a 4 point Likert-type scale, coded from 0 - 10 for conversion into continuous variables (None = 0; Mild = 1 - 3; Moderate = 4 - 6 ; Severe = 7 - 10).
Straining | Assessed daily throughout both dietary protocols (7 days for each dietary protocol)
  Straining will be recorded daily in a symptom diary and measured using a 4 point Likert-type scale, coded from 0 - 10 for conversion into continuous variables (None = 0; Mild = 1 - 3; Moderate = 4 - 6 ; Severe = 7 - 10).
Incomplete Defecation | Assessed daily throughout both dietary protocols (7 days for each dietary protocol)
  Incomplete defection will be recorded daily in a symptom diary and measured using a 4 point Likert-type scale, coded from 0 - 10 for conversion into continuous variables (None = 0; Mild = 1 - 3; Moderate = 4 - 6 ; Severe = 7 - 10).
Stool Form | Assessed daily throughout both dietary protocols (7 days for each dietary protocol)
  Stool form will be measured using the Bristol Stool Form Scale. Type 1 - Separate hard lumps, like nuts (hard to pass), Type 2 - Sausage shaped, but lumpy, Type 3 - Like a sausage but with cracks on its surface, Type 4 - Like a sausage or snake, smooth and soft, Type 5 - Soft blobs with clear cut edges (passed easily), Type 6 - Fluffy pieces with ragged edges, a mushy stool, and Type 7 - Watery, no solid pieces, entirely liquid. Stool Types 1 and 2 are associated with constipation, while stool Types 5 - 7 are associated with diarrhoea. Stool Types 3 and 4 are considered normal stools.
Frequency of defecation | Assessed daily throughout both dietary protocols (7 days for each dietary protocol)
  Frequency of defecation will be recorded daily in a symptom diary.

SECONDARY OUTCOMES:
Fatigue | Assessed on the last day of both dietary protocols (Day 7 of each dietary protocol)
  Fatigue will be recorded and measured using the Fatigue Assessment Scale (FAS) (Michielsen et al., 2003), using a 5 point Likert-type scale, coded from 1 - 5 for conversion into continuous variables (None = 1; Sometimes = 2; Regularly = 3; Often = 4; Always = 5). Question 1 - I am bothered by fatigue; Question 2 - I get tired very quickly; Question 3 - I don't do much during the day; Question 4 - I have enough energy for everyday life; Question 5 - Physically, I feel exhausted; Question 6 - I have problems starting things; Question 7 - I have problems thinking clearly; Question 8 - I feel no desire to do anything; Question 9 - Mentally, I feel exhausted and Question 10 - When I am doing something, I can concentrate quite well. Question 4 and 10 are to be reverse scored. Total scores can range from 10, indicating the lowest level of fatigue, to 50, denoting the highest.
Mental Fatigue | Assessed on the last day of both dietary protocols (Day 7 of each dietary protocol)
  Mental fatigue will be measured using the Fatigue Assessment Scale (FAS), using a 5 point Likert-type scale, coded from 1 - 5 for conversion into continuous variables (None = 1; Sometimes = 2; Regularly = 3; Often = 4; Always = 5). Only questions 6 - 10 will be used to calculate the mental fatigue score. Question 6 - I have problems starting things; Question 7 - I have problems thinking clearly; Question 8 - I feel no desire to do anything; Question 9 - Mentally, I feel exhausted and Question 10 - When I am doing something, I can concentrate quite well. Question 10 is to be reverse scored. Total scores can range from 5, indicating the lowest level of fatigue, to 25, denoting the highest.
Physical Fatigue | Assessed on the last day of both dietary protocols (Day 7 of each dietary protocol)
  Physical fatigue will be measured using the Fatigue Assessment Scale (FAS), using a 5 point Likert-type scale, coded from 1 - 5 for conversion into continuous variables (None = 1; Sometimes = 2; Regularly = 3; Often = 4; Always = 5). Only questions 1 - 5 will be used to calculate the mental fatigue score. Question 1 - I am bothered by fatigue; Question 2 - I get tired very quickly; Question 3 - I don't do much during the day; Question 4 - I have enough energy for everyday life; Question 5 - Physically, I feel exhausted. Question 4 is to be reverse scored. Total scores can range from 5, indicating the lowest level of fatigue, to 25, denoting the highest.

CONTACTS AND LOCATIONS:
Overall Officials: Camilla Bunn, Principal Investigator — University of Suffolk
Locations (1):
- University of Suffolk, Ipswich, Suffolk, United Kingdom

REFERENCES:
- [Background] Ibrahim F, Stribling P. A 5Ad Dietary Protocol for Functional Bowel Disorders. Nutrients. 2019 Aug 17;11(8):1938. doi: 10.3390/nu11081938. PMID 31426496
- [Background] Ibrahim F, Stribling P. Reply to "A Gluten Reduction Is the Patients' Choice for a Dietary 'Bottom Up' Approach in IBS-A Comment on "A 5Ad Dietary Protocol for Functional Bowel Disorders" Nutrients 2019, 11, 1938". Nutrients. 2020 Jan 3;12(1):140. doi: 10.3390/nu12010140. PMID 31947828
- [Background] Gibson PR, Shepherd SJ. Personal view: food for thought--western lifestyle and susceptibility to Crohn's disease. The FODMAP hypothesis. Aliment Pharmacol Ther. 2005 Jun 15;21(12):1399-409. doi: 10.1111/j.1365-2036.2005.02506.x. PMID 15948806
- [Background] Lewis SJ, Heaton KW. Stool form scale as a useful guide to intestinal transit time. Scand J Gastroenterol. 1997 Sep;32(9):920-4. doi: 10.3109/00365529709011203. PMID 9299672
- [Background] Michielsen HJ, De Vries J, Van Heck GL. Psychometric qualities of a brief self-rated fatigue measure: The Fatigue Assessment Scale. J Psychosom Res. 2003 Apr;54(4):345-52. doi: 10.1016/s0022-3999(02)00392-6. PMID 12670612